CLINICAL TRIAL: NCT02181686
Title: Iperia Family / Sentus QP Master Study
Brief Title: Iperia/Sentus QP Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Heart Failure; Tachyarrhythmia
Keywords: Heart Failure; Iperia ICD family; Sentus QP left ventricular lead; Quadripolar CRT-D system
MeSH Terms: conditions — Heart Failure; Tachycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sentus QP group: Patients with standard indication for CRT-D therapy who will be implanted with Sentus QP LV lead and the BIOTRONIK HF-T QP device.
- VR-T/DR-T group: Patients with standard indication for ICD therapy who will be implanted with either single chamber ICD or dual chamber ICD of the Iperia ICD family

SUMMARY:
The objective of this study is to confirm the safety and efficacy of the new Sentus OTW QP LV lead and Iperia ICD family. The study focuses on the safety and efficacy of the QP device system.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to understand the nature of the study and provides written informed consent.
* Patient meets a standard indication for CRT-D (Sentus QP group) or ICD therapy.
* Patient is able and willing to complete the planned follow-up visits at the investigational site.
* Patient accepts the Home Monitoring® concept.
* Age is ≥ 18 years.
* Sentus QP group only: Patient is a candidate for a new (de novo) implant or an upgrade from an existing ICD or pacemaker utilizing a BIOTRONIK Sentus QP lead

Exclusion Criteria:

* Patient has a standard contraindication for CRT-D (Sentus QP group) or ICD therapy.
* Sentus QP group only: Currently implanted with an endocardial or epicardial LV lead or had prior attempt to place a LV lead.
* Sentus QP group only: Cardiac surgery procedure (coronary bypass graft, valve surgery, or ablation) that is planned to occur within 3 months after implantation.
* Patient is expected to receive ventricular assist device or heart transplantation within the next 3 months.
* Patient is pregnant or breastfeeding.
* Life expectancy of less than 3 months
* Participating in another cardiac clinical investigation with active treatment arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient collective consists mainly of heart failure patients with CRT-D indication according to current guidelines. In addition 50 patients with an indication for single or dual chamber ICD will be enrolled in the study. The investigator will select patients who are appropriate for particiation from his general patient population.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Sentus QP LV lead: Serious Adverse Device Effect (SADE) free rate | 3 months
  The safety of the LV lead will be evaluated by asking the investigator to record any adverse event. While all adverse events have to be recorded throughout the study, only the number of SADEs possibly or securely related to the LV lead will be the basis for endpoint calculation of the SADE-free rate.
Iperia ICD family: SADE free rate | 3 months
  The safety of the Iperia ICD family will be evaluated by asking the investigator to record any adverse event. While all adverse events have to be recorded throughout the study, only the number of SADEs possibly or securely related to the pacemaker will be the basis for endpoint calculation of the SADE-free rate.

SECONDARY OUTCOMES:
LV pacing threshold | 3 months
  Lv pacing threshold measured in the final programmed pacing vector

OTHER OUTCOMES:
Collection of data of interest: Handling of LV lead during implantation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Werner Jung, Prof. Dr., Principal Investigator — Schwarzwald-Baar Klinikum Villingen-Schwenningen, Germany
Locations (24):
- Landesklinikum, Sankt Pölten, Austria
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense
  - Aarhus University Hospital, Skejby
- Jyväskylä Central Hospital, Jyväskylä, Finland
- Germany (9):
  - Herz- und Diabetes Zentrum, Bad Oeynhausen
  - SRH Wald-Klinikum, Gera
  - Medizinische Hochschule Hannover, Hanover
  - UKSH Campus Lübeck, Lübeck
  - Märkische Kliniken Lüdenscheid, Lüdenscheid
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinikum München-Bogenhausen, Munich
  - Johanniter Krankenhaus, Stendal
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
- Ospedale Pugliese Ciaccio, Catanzaro, Italy
- Paul Stradins Clinical University Hospital, Riga, Latvia
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Isala Klinieken, Zwolle
- National Heart Centre, Singapore, Singapore
- Hospital Clinic de Barcelona, Barcelona, Spain
- Switzerland (3):
  - Kantonsspital Lucerne, Lucerne
  - Cardiocentro Ticino, Lugano
  - Triemlispital Zurich, Zurich
- Russels Hall Hospital, Brighton, United Kingdom